CLINICAL TRIAL: NCT02218957
Title: Restrictive Extended Pouch in Roux-en-Y Gastric Bypass: a Prospective Randomized Control Trial
Brief Title: Extended Pouch Roux-en-Y Gastric Bypass Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ExtPouch
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Morbid Obesity
Keywords: Bariatric surgery; Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard RYGB (Active Comparator): Standard RYGB
  Interventions: Procedure: Standard RYGB
- Extended Pouch RYGB (Experimental): Restrictive/extended pouch RYGB
  Interventions: Procedure: Extended Pouch RYGB

INTERVENTIONS:
Procedure: Extended Pouch RYGB
  Arms: Extended Pouch RYGB
Procedure: Standard RYGB
  Arms: Standard RYGB

SUMMARY:
Morbid obesity is an increasing medical problem in the western countries. It's related to comorbidities as diabetes mellitus, hypertension, OSAS, arthrosis and hypercholesterolemia. The Roux-en-Y Gastric Bypass (RYGB) is an effective surgical therapy for morbidly obese patients. A part of these patients will have disappointing results, and have weight regain on the long term. Some studies show more weight reduction by increasing the biliopancreatic limb in patients with morbid obesity.

The objective of this study is to investigate the effect of a restrictive/extended pouch on weight reduction in morbidly obese patients undergoing RYGB-surgery. We hypothesize that the restrictive/extended pouch results in more weight reduction.

The study design is a prospective, randomized control trial. The patients will be randomized in 2 groups: a standard RYGB (normal pouch) and restrictive/extended pouch RYGB.

ELIGIBILITY:
Inclusion Criteria:

Patient eligible for bariatric surgery according Fried guidelines

Primary Gastric bypass

* BMI 35 - 40 with a comorbidity
* or BMI > 40

Exclusion Criteria:

* Exclusion criteria for bariatric surgery (Fried Guidelines)
* Patients with language problems that interveins to follow medical advises
* Genetic diseases that intervens to follow medical advises
* Chronic bowel diseases
* Nephrologic (MDRD <30) of liver diseases (AST/ALT more than twice the norm)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Weight reduction | 2 years
  Excess weight loss (%EWL)

SECONDARY OUTCOMES:
Change in comorbidities | 2 years
  Preoperatively the number of patients with comorbidities will be calculated. At two year follow-up this will be calculated again. Patients will be divided in groups:
  1. comorbidity resolved
  2. comorbidity improved
  3. comorbidity unchanged
  4. comorbidity worsened
  This will be done for diabetes mellitus, hypertension, dyslipidemia and OSAS.
Change in comorbidities | 2 years
  Preoperatively the number of patients with comorbidities will be calculated. At two year follow-up this will be calculated again. Patients will be divided in groups:
  1. comorbidity resolved
  2. comorbidity improved
  3. comorbidity unchanged
  4. comorbidity worsened
  This will be done for diabetes mellitus, hypertension, dislipidemia and OSAS.

OTHER OUTCOMES:
Complications | 2 years
  Complications will be divided in short-term complications (within 30 days after operation) and long-term complications (after 30 days). All adverse event will be registered.
Quality of life | 2 years
  The quality of life will be assessed by using the BAROS.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Homan, MD, Principal Investigator — Rijnstate Hospital Arnhem
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands